CLINICAL TRIAL: NCT04785209
Title: Mean Platelet Volume and STEMI Clinical Risk Scores in Prediction of Impaired Myocardial Perfusion In Acute STEMI Patients Undergoing PPCI.
Brief Title: Mean Platelet Volume and STEMI Clinical Risk Scores in Prediction of Impaired Myocardial Perfusion In Acute STEMI Patients Undergoing Primary Percutaneous Coronary Intervention.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Reymon Sadik Salama, Principle invistigator, Assiut University
Other Study IDs: Prediction of No reflow
Record Dates: First submitted 2020-09-23; First posted 2021-03-05 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: No-Reflow Phenomenon
MeSH Terms: conditions — No-Reflow Phenomenon | interventions — Mean Platelet Volume; Lymphocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No complication: Thrombolysis in myocardial infarction flow grade III flow after PPCI, mean platelet volume, lymphocyte ratio, detailed echo within 24 hrs of admission, clinical STEMI risk scores
  Interventions: Other: Mean platelet volume, lymphocyte number, STEMI clinical risk scores
- No reflow: No reflow phenomenon after pci on STEMI patients, mean platelet volume, lymphocyte ratio, detailed echo within 24 hrs of admission, clinical STEMI risk scores
  Interventions: Other: Mean platelet volume, lymphocyte number, STEMI clinical risk scores

INTERVENTIONS:
Other: Mean platelet volume, lymphocyte number, STEMI clinical risk scores — Lab parameters

SUMMARY:
Predicting no reflow in ppci of STEMI patients using mean platelet volume together with STEMI clinical risk scores

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with acute STEMI, within 24 hours of symptoms, fulfilling criteria for PPCI protocol in our facility

Exclusion Criteria:

* patients presenting more than 24 hours of symptoms onset
* patients not eligible for PPCI program in our facility

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All STEMI patients presenting within 24 hrs of onset of symptoms
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participents with No reflow after PPCI and in hospital mortality | Within 48 hours from admission
  No reflow: suboptimal myocardial reperfusion through a part of coronary circulation without angiographic evidence of mechanical vessel obstruction.
  In hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Shams elddin, Professor, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt